CLINICAL TRIAL: NCT01342887
Title: Cyclosporine Modulation of Drug Resistance in Combination With Pravastatin, Mitoxantrone, and Etoposide for Adult Patients With Relapsed/Refractory Acute Myeloid Leukemia (AML): A Phase 1/2 Study
Brief Title: Cyclosporine, Pravastatin Sodium, Etoposide, and Mitoxantrone Hydrochloride in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Roland Walter, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2409.00; NCI-2011-00657 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-04-22; First posted 2011-04-27 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Cyclosporine; Pravastatin; Mitoxantrone; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (immunosuppression, enzyme inhibitor, and chemo) (Experimental): Patients receive cyclosporine IV continuously on days 5-9. Patients also receive pravastatin sodium PO every 6 hours on days 1-10, etoposide IV continuously on days 5-9, and mitoxantrone hydrochloride IV continuously on days 5-9. Treatment repeats for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients achieving CR/CRi may receive 2 additional courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cyclosporine; Drug: pravastatin sodium; Drug: mitoxantrone hydrochloride; Drug: etoposide; Procedure: bone marrow aspiration

INTERVENTIONS:
Drug: cyclosporine — Given IV
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Drug: pravastatin sodium — Given PO
  Other Names: PRAV; Pravachol
Drug: mitoxantrone hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Novantrone
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Procedure: bone marrow aspiration — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of etoposide and mitoxantrone hydrochloride when given together with cyclosporine and pravastatin sodium and to see how well they work in treating patients with relapsed or refractory acute myeloid leukemia (AML). Cyclosporine may inhibit efflux of cancer drugs out of cancer cells and may thereby improve chemotherapy treatment for AML. Pravastatin sodium may stop the growth of cancer cells by blocking some of the nutrients needed for cell growth. Drugs used in chemotherapy, such as etoposide and mitoxantrone hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving cyclosporine together with pravastatin sodium, etoposide, and mitoxantrone hydrochloride may kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated doses of mitoxantrone (mitoxantrone hydrochloride) and etoposide in combination with pravastatin (pravastatin sodium) and cyclosporine.

SECONDARY OBJECTIVES:

I. Describe the complete remission (CR)/CR with incomplete peripheral blood count recovery (CRi) rate after up to 2 cycles of induction therapy.

II. Describe the disease-free survival of patients that achieve CR/CRi. III. Estimate the frequency and severity of regimen-associated toxicities, along with 28-day mortality after start of study treatment.

OUTLINE: This is a phase I/II, dose-escalation study of etoposide and mitoxantrone hydrochloride in combination with pravastatin sodium and cyclosporine.

Patients receive cyclosporine intravenously (IV) continuously on days 5-9. Patients also receive pravastatin sodium orally (PO) every 6 hours on days 1-10, etoposide IV continuously on days 5-9, and mitoxantrone hydrochloride IV continuously on days 5-9. Treatment repeats for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients achieving CR/CRi may receive 2 additional courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-related mortality (TRM) score =< 9.2 as calculated with simplified model
* Prior morphological diagnosis of AML according to the 2008 World Health Organization (WHO) diagnostic criteria; patients with biphenotypic AML are eligible; patients with acute promyelocytic leukemia with t(15;17)(q22;q12) and variants are ineligible
* Relapsed/persistent disease as defined by International Working Group criteria; outside diagnostic material is acceptable as long as peripheral blood and/or bone marrow slides are reviewed at the study institution; flow cytometric analysis of peripheral blood and/or bone marrow should be performed according to institutional practice guidelines
* Patients with prior autologous or allogeneic hematopoietic cell transplantation (HCT) are eligible if relapse occurs > 180 days post-transplant provided symptoms of graft-versus host disease are well controlled with stable use of immunosuppressive agents
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-3, assessed at time of registration
* Should be off any active therapy for AML with the exception of hydroxyurea or low-dose cytarabine (=< 100 mg/m^2) for at least 14 days prior to study registration unless patient has rapidly progressive disease, and all Grade 2-4 non-hematologic toxicities must have resolved
* Bilirubin =< 2 x Institutional Upper Limit of Normal (IULN) unless elevation is thought to be due to hepatic infiltration by AML, Gilbert's syndrome, or hemolysis (assessed within 7 days prior to registration)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamic pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2 x IULN unless elevation is thought to be due to hepatic infiltration by AML (assessed within 7 days prior to registration)
* Serum creatinine =< 1.5 x IULN (assessed within 7 days prior to registration)
* Left ventricular ejection fraction >= 40%, assessed within 28 days prior to registration, e.g. by multi gated acquisition scan (MUGA) scan or echocardiography, or other appropriate diagnostic modality, and no clinical evidence of congestive heart failure; if the patient had anthracycline-based therapy since the most recent cardiac assessment, cardiac evaluation should be repeated if there is clinical or radiographical suspicion of cardiac dysfunction, or if the previous cardiac assessment was abnormal
* Patients with symptoms/signs of hyperleukocytosis or white blood cell (WBC) > 100,000/uL can be treated with leukapheresis prior to enrollment
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Ability to understand and the willingness to sign a written informed consent document; the consent can be obtained from a legally authorized representative if the patient is unable to provide informed consent

Exclusion Criteria:

* Diagnosis of another malignancy, unless the patient was diagnosed at least 2 years earlier and has been disease-free for at least 6 months following the completion of curative intent therapy with the following exceptions:

  * Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed
  * Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed
* Refractory/relapsing blast crisis of chronic myelogenous leukemia (CML)
* Known hypersensitivity to any study drug
* Human immunodeficiency virus (HIV)-positive patients are excluded if their cluster of differentiation (CD)4 count is below 200 cells/uL or if they have active acquired immune deficiency syndrome (AIDS)-related complications, as these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy
* Pregnancy or lactation; women of childbearing potential must undergo pregnancy test within 7 days prior to registration
* Uncontrolled systemic fungal, bacterial, viral, or other infection (defined as exhibiting progressive signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
* Patients may not be receiving any other investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roland Walter, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Immunosuppression, Enzyme Inhibitor, and Chemo)
Started | 6
Completed | 4
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Immunosuppression, Enzyme Inhibitor, and Chemo)
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 51 [40 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Doses Mitoxantrone Hydrochloride and Etoposide When Combined With Cyclosporine and Pravastatin Sodium
Description: Determine the doses of mitoxantrone and etoposide that, when combined with CSA and pravastatin, meet minimum standards for both efficacy and toxicity and have the highest efficacy rate among several mitoxantrone and etoposide doses.
  Assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: After completion of first 2 courses, up to 22 weeks
Measure: Number; unit: doses tolerated
Arm/Group | Treatment (Immunosuppression, Enzyme Inhibitor, and Chemo)
Number analyzed (Participants) | 6
doses tolerated | 0

2. Secondary Outcome: CR/CRi
Description: Describe the disease-free survival of patients that achieve Complete Remission (CR)/CR with inadequate recovery of peripheral blood cell counts (CRi).
  Categorized according to criteria recommended by an International Working Group.
Time Frame: After completion of first 2 courses, up to 22 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Immunosuppression, Enzyme Inhibitor, and Chemo)
Number analyzed (Participants) | 6
Participants
  CR | 0
  CRi | 0
  CR/CRi not achieved | 6

3. Secondary Outcome: Disease-free Survival of Patients That Achieve CR/CRi
Description: Describe the disease-free survival of patients that achieve CR/CRi.
Time Frame: Up to 4.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Immunosuppression, Enzyme Inhibitor, and Chemo)
Number analyzed (Participants) | 6
Participants
  0-6month survival of those achieving CR/CRi | 0
  >6month survival of those achieving CR/CRi | 0
  Participants who do not achieve CR/CRi | 6

4. Secondary Outcome: Frequency and Severity of Regimen-associated Toxicities
Description: Estimate the frequency and severity of regimen-associated toxicities, along with 28-day mortality after start of study treatment
Time Frame: At 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Immunosuppression, Enzyme Inhibitor, and Chemo)
Number analyzed (Participants) | 6
Participants
  Early death (within 28 days) | 2
  Experienced Dose-Limiting Toxicity | 1
  Persistent Disease | 3

ADVERSE EVENTS:
Arm/Group | Treatment (Immunosuppression, Enzyme Inhibitor, and Chemo)
Serious Adverse Events (participants affected / at risk) | 5/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Immunosuppression, Enzyme Inhibitor, and Chemo) (N=6)
Sepsis (Infections and infestations) | 4 (4)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Immunosuppression, Enzyme Inhibitor, and Chemo) (N=6)
Acute Kidney Injury (Renal and urinary disorders) | 3 (4)
Acute toxic-metabolic encephalopathy (Nervous system disorders) | 1 (1)
Altered Mental Status (Psychiatric disorders) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anuria (Renal and urinary disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blanched buttocks (Skin and subcutaneous tissue disorders) | 1 (1)
Bronchospasms (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Burning sensation during urination (Renal and urinary disorders) | 1 (1)
Burning sensation during infusion (Injury, poisoning and procedural complications) | 3 (3)
Cellulitis (Infections and infestations) | 1 (1)
Chest pain (General disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Coagulase Negative Staphylococcus Bacteremia (Infections and infestations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Dizziness (Nervous system disorders) | 2 (2)
E. Coli Urinary Tract Infection (Infections and infestations) | 1 (1)
Ear pain to palpitation (Ear and labyrinth disorders) | 1 (1)
Periobital Edema (Skin and subcutaneous tissue disorders) | 2 (2)
Transaminitis (Hepatobiliary disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 5 (5)
Febrile nonhemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1 (1)
Scalp rash (Skin and subcutaneous tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Heartburn (Gastrointestinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2)
Hypertension (Vascular disorders) | 6 (6)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Hypothermia (General disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Jaundice (Investigations) | 1 (1)
Leg Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Leukemia cutis (Skin and subcutaneous tissue disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 6 (7)
Malaise (General disorders) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 6 (6)
Multifocal pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (6)
Nervousness/agitation (Psychiatric disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 (7)
Oral Thrush (Gastrointestinal disorders) | 1 (1)
Pain on left areola, superficial (Reproductive system and breast disorders) | 1 (1)
Pain, right axillary area (Skin and subcutaneous tissue disorders) | 2 (2)
Palpitation (Cardiac disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 3 (3)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary Aspergillosis (Immune system disorders) | 1 (1)
Rash, chest (Infections and infestations) | 3 (3)
Restlessness (Nervous system disorders) | 1 (1)
Rhabdomyolysis (Renal and urinary disorders) | 1 (1)
Rhinovirus (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sinus Infection (Infections and infestations) | 1 (1)
Tachycardia (Cardiac disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema, bilateral hand and feet (General disorders) | 2 (2)
Edema, face (General disorders) | 1 (1)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tremors (Nervous system disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Vancomycin-Resistant Enterococci Bacteremia (Infections and infestations) | 2 (2)
Viral upper respiratory infection (Infections and infestations) | 1 (1)
Volume Retention (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
Weight Gain (Investigations) | 1 (1)
Withdrawn/Unwilling to communicate (Psychiatric disorders) | 1 (1)
Extraocular muscle paresis, worsening (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes